CLINICAL TRIAL: NCT06433960
Title: A Cross-Sectional Study and a Novel Screening Survey for Radial Artery Assessment in Surgical Coronary Revascularisation
Brief Title: Radial Artery Assessment in Surgical Coronary Revascularisation
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 24/SC/0076
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Bypass Grafting; Coronary Artery Disease
Keywords: Radial Artery; Modified Allen Test; Barbeau Test; Ultrasonography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiovascular sample group: Cardiac patients undergoing elective or urgent coronary artery bypass graft surgery and radial artery harvest in two Cardiothoracic hospitals.
  Interventions: Diagnostic Test: Modified Allen Test; Diagnostic Test: Pulse-oximetry guided Modified Allen Test; Diagnostic Test: Barbeau Test; Diagnostic Test: Ultrasound examination of the forearm arteries; Diagnostic Test: Measurement of oxygen saturation; Other: Radial Artery Quality Evaluation Survey; Other: Follow-up Radial Artery Harvesting Scale

INTERVENTIONS:
Diagnostic Test: Modified Allen Test — Pre-operative intervention aimed at evaluating if forearm blood vessels (ulnar artery and collateral) would supply an adequate blood flow to the arm if the radial artery was harvested. Duration: 1 minute.
  Instruct the patient to clench their wrist while the examiner occlude with three fingers the patients ulnar and radial arteries; instruct the patient to unclench their wrist; release the ulnar artery. The MAT result is negative or positive considering in how long the palm flushes:
  ≤5 seconds: negative MAT; good collateral hand circulation (suggesting harvestable radial artery).
  greater than 5 seconds: positive MAT; poor collateral hand circulation (suggesting not-harvestable radial artery).
Diagnostic Test: Pulse-oximetry guided Modified Allen Test — Pre-operative intervention aimed at evaluating if forearm blood vessels (ulnar artery and collateral) would supply an adequate blood flow to the arm if the radial artery was harvested. Duration: 1 minute.
  A pulse-oximetry probe is positioned on the patients index finger; both radial and ulnar arteries are occluded by the examiner (with three fingers) until flattening of pulse waveform is obtained. Pressure on the ulnar artery is released and the result of the assessment is calculated considering in how long the pulse waveform returns to baseline:
  ≤5 seconds: negative result (suggesting harvestable radial artery). greater than 5 seconds: positive result (suggesting not harvestable radial artery).
  (Busti and Kellogg, 2015)
Diagnostic Test: Barbeau Test — Pre-operative intervention aimed at evaluating if forearm blood vessels (ulnar artery and collateral) would supply an adequate blood flow to the arm if the radial artery was harvested. Duration: 2 minutes.
  A pulse-oximetry probe is positioned on the patients thumb; the radial artery is then compressed by the examiner, and the pulse waveform is analysed for up to 120 seconds, providing four result patterns of ulno-palmar patency:
  1. No damping of the pulse tracing immediately after compression (suggesting harvestable radial artery)
  2. Damping of the pulse tracing (suggesting harvestable radial artery)
  3. Loss of the pulse tracing, followed by recovery within 120 sec (suggesting harvestable radial artery)
  4. Loss of the pulse tracing, without recovery within 120 sec (suggesting not harvestable radial artery).
  (Zalocar et al., 2020)
Diagnostic Test: Ultrasound examination of the forearm arteries — Pre-operative intervention aimed at evaluating morphological characteristics (diameter, presence of calcifications) of the radial and ulnar arteries. Duration: 5 minutes.
  The radial artery is surgically exposed (negative result) when the following apply:
  1. ulnar artery inner diameter ≥2 mm
  2. radial artery inner diameter ≥2 mm
  3. absence of radial artery intraluminal calcifications and plaques.
  (Vukovic et al., 2017)
Diagnostic Test: Measurement of oxygen saturation — Intra-operative intervention aimed at evaluating the blood oxygen level in the hand if the radial artery was harvested. Duration: 1 minute.
  The radial artery is surgically harvested when the oxygen saturation reading (SpO2) from the thumb through pulse-oximetry remains at 95% or above when an occlusive atraumatic clamp is applied on the mobilised radial artery.
Other: Radial Artery Quality Evaluation Survey — Intra-operative intervention (validated structured questionnaire) aimed at evaluating anatomical and physiological characteristics of the radial artery and suitability for coronary graft implantation.
  The radial artery is surgically harvested when its morphology and pathology (diameter, calcifications, presence of pulsatile flow), quality of harvesting technique and surgical accessibility are considered satisfactory, good or optimal.
  The Radial Artery Quality Evaluation Survey is completed by surgical care practitioners.
Other: Follow-up Radial Artery Harvesting Scale — Postoperative intervention (ordinal symptoms scale) aimed at evaluating patients finger movements, cold tolerance sensitivity and tactile/touch perception at post-operative day 2 to 5 and at follow-up appointment (3-6 weeks after surgery). Bilateral comparison between hands and forearms is undertaken. Tactile perception is assessed through monofilaments (single touch). Cold sensitivity is assessed through the use of ice-pack.
  The Follow-up Radial Artery Harvesting Scale was developed from a verbal rating scale (VRS) questionnaire documented in the literature. The VRS questionnaire was re-adapted to appreciate people postoperative experience with their finger movements, cold sensitivity and tactile/touch perception of their forearm.

SUMMARY:
The goal of this observational study is to learn about how screening tests inform the radial artery (RA) suitability for harvesting and coronary bypass grafting in adults with ischaemic heart disease. The main question it aims to answer is:

• What factors influence the diagnostic accuracy of RA screening in patients undergoing surgical coronary revascularisation?

Participants will:

* Receive an assessment of their RA through routinely used techniques (Modified Allen Test +/- pulse-oximetry, Barbeau Test and Ultrasound examination)
* Answer a symptoms scale about their physical experience after surgery

DETAILED DESCRIPTION:
A multi-centre cross-sectional study design to investigate the validity of radial artery (RA) assessment techniques in adults with ischaemic heart disease undergoing surgical coronary revascularisation with their RA being selected as an autologous graft conduit.

Patients taking part in the study will receive an assessment of the arterial forearm circulation from their non-dominant upper extremity through multiple observations.

Pre-operative observations. Before surgery (in the ward environment after the patient is being admitted or whilst patient in the anaesthetic room) the forearm blood circulation is measured through a Modified Allen Test (MAT) (+/- pulse-oximetry), Barbeau Test and Ultrasonography examination. Assessment will be performed by experienced Surgical Care Practitioners/Advanced Nurse Practitioners/Cardiac Specialist Registrars. These assessments will inform the decision to surgically expose the RA.

Intra-operative observations. Oxygen saturation readings are taken prior to harvest the RA. Once the RA is surgically harvested a series of measures are taken through a validated structured questionnaire: the Radial Artery Quality Evaluation Survey (RAQES).

Observations at 4-6 weeks post operation. Patients finger movements, cold tolerance sensitivity and tactile/touch perception is measured through an ordinal symptoms scale (Follow-up Radial Artery Harvesting Scale) at post-operative day 2-5 and at follow-up appointment (3-6 weeks after surgery). Bilateral comparison between hands and forearms will be undertaken. A Surgical Care Practitioner will perform this assessment post-operatively.

Consecutive sampling will be used for the recruitment of study participants. The minimum required number of participants to test and verify research hypotheses is sixty-nine patients (N=69). An adaptive trial design will be implemented: at quarterly assessment points the statistical power is assessed and the remaining sample size required is updated accordingly.

Sample size calculation was undertaken using G*Power software (version 3.1) using Chi-squared Test and adopting optimal effect size (w=0.4) and power (0.8).

Descriptive and inferential statistics will be used to perform quantitative analyses. Descriptive statistics (mode, median) will be implemented to analyse RAQES answers and ordinal symptoms scale findings and cross-tabulation used to record relationship between variables. Data analysis will also include measurement of sensitivity, specificity, positive and negative predictive values to investigate the validity of the RA assessment techniques. Correlational analysis will be implemented and Receiver Operating Characteristic curve analysis will be used to compare the diagnostic accuracy of the MAT, pulse-oximetry guided MAT and Barbeau Test with the ultrasonography examination.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults patients undergoing elective or urgent coronary artery bypass graft (CABG) surgery and radial artery (RA) harvesting in two Cardiothoracic hospitals.

Exclusion Criteria:

* Paediatric patients and/or adult patients undergoing emergency CABG will not be considered within the participants of this cross-sectional study, as well as patients lacking capacity to consent and non-English speaking patients requiring use of interpreters. Patients not wishing to participate in the study will also not be recruited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with ischaemic heart disease undergoing coronary bypass surgery and radial artery harvest at Royal Papworth and Royal Brompton hospitals will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Radial Artery Assessment Techniques | From enrollment to the end of treatment at 12 weeks.
  Measure the sensitivity of the Modified Allen test (+/- pulse-oximetry), the Barbeau Test and ultrasonography examination.
Specificity of Radial Artery Assessment Techniques | From enrollment to the end of treatment at 12 weeks.
  Measure the specificity of the Modified Allen test (+/- pulse-oximetry), the Barbeau Test and ultrasonography examination.
Negative and Positive predictive values of Radial Artery Assessment Techniques | From enrollment to the end of treatment at 12 weeks.
  Measure the negative and positive predictive values of the Modified Allen test (+/- pulse-oximetry), the Barbeau Test and ultrasonography examination.

SECONDARY OUTCOMES:
Radial Artery Quality Evaluation | From enrollment to surgical harvesting of the radial artery at day 1-2 after hospitalisation.
  Measure the morphological and physiological quality of radial arteries through a validated structured questionnaire (Radial Artery Quality Evaluation Survey)
Patients Physical Experience Evaluation | From day of surgery to the end of treatment at 12 weeks.
  Measure the patients' finger movements, cold tolerance sensitivity and tactile/touch perception through an ordinal symptoms scale (Follow-up Radial Artery Harvesting Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo De Franco, MSc SCP, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London, England
  - Royal Papworth Hospital, Cambridge, England/Cambridgeshire

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. Shared IPD will be presented in a de-identified (anonymised) format for each participant and will include information about interventions or tests received and outcomes observed.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 3 years after the publication of results.
Access Criteria: Researchers wishing to conduct a diagnostic accuracy analysis of the tests (interventions) under investigation car require copy of the anonymised IPD and supporting information to the principal investigator.
  A proposal describing the planned analysis must be provided and a data sharing agreement form (requested to the sponsoring institution) must be signed.
  Further instructions for obtaining access are available at the link below:
  https://royalpapworth.nhs.uk/research-and-development or contacting: papworth.randdadmin@nhs.net
URL: https://royalpapworth.nhs.uk/research-and-development

REFERENCES:
- [Background] Zalocar LAD, Doroszuk G, Goland J. Transradial approach and its variations for neurointerventional procedures: Literature review. Surg Neurol Int. 2020 Aug 15;11:248. doi: 10.25259/SNI_366_2020. eCollection 2020. PMID 32905334
- [Background] Vukovic P, Peric M, Radak S, Aleksic N, Unic-Stojanovic D, Micovic S, Stojanovic I, Milojevic P. Preoperative Insight Into the Quality of Radial Artery Grafts. Angiology. 2017 Oct;68(9):790-794. doi: 10.1177/0003319716686014. Epub 2017 Jan 5. PMID 28056520
- See also: Busti, A.J. and Kellogg, D. (2015) Allens Test. — https://www.ebmconsult.com/articles/physica-exam-allens-test
- See also: Kinoue, T. and Arai, M. (2021) Comparison of Rating Scale Methods for Cold Sensation in Kampo Medicine, International Medical Journal, 28(1), pp.94-97. — https://seronjihou.files.wordpress.com/2021/05/281094.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT06433960/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT06433960/ICF_002.pdf